CLINICAL TRIAL: NCT04139590
Title: The Evaluation of Smartphone Versions of the Visual Analogue Scale and Numeric Rating Scale as Postoperative Pain Assessment Tools
Brief Title: Evaluation of Smartphone Versions of VAS and NRS for Use in Adults
Acronym: Panda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Children's Hospital (Other); Providence Health & Services (Other)
Responsible Party: Principal Investigator, Ron Ree, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H1601196
Record Dates: First submitted 2018-04-30; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; Visual Analogue Scale; Numeric Rating Scale; Smartphone
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants had to use versions of the scale. They were randomized to using Panda or the original version of the scales first. Scores obtained using the two versions are then compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Visual Analogue Scale - Original (Placebo Comparator): Participants indicated the intensity of their pain by marking a "X" along the original paper version of the Visual Analogue Scale.
  Interventions: Device: Visual Analogue Scale - Original
- Visual Analogue Scale - Panda (Active Comparator): Participants indicated the intensity of their pain by marking a "X" on the smartphone screen using the Panda of the Visual Analogue Scale.
  Interventions: Device: Panda
- Numeric Rating Scale - Original (Placebo Comparator): Participants indicated the intensity of their pain by marking a "X" along the original paper version of the Numeric Rating Scale.
  Interventions: Device: Visual Analogue Scale - Original
- Numeric Rating Scale - Panda (Active Comparator): Participants indicated the intensity of their pain by marking a "X" on the smartphone screen using the Panda of the Numeric Rating Scale.
  Interventions: Device: Panda

INTERVENTIONS:
Device: Panda
  Arms: Numeric Rating Scale - Panda; Visual Analogue Scale - Panda
Device: Visual Analogue Scale - Original
  Arms: Numeric Rating Scale - Original; Visual Analogue Scale - Original

SUMMARY:
A large number of patients experience significant pain after surgery, and more patients report pain after discharge from hospital than before. This issue has been observed in patients who receive peripheral nerve blocks, the effects of which often wear off after discharge. There are numerous barriers to the effective control of pain away from the direct supervision of medical professionals, and personalized management strategies are necessary in order to overcome these barriers. The first step of adequate pain management is accurate pain assessment. Therefore, this study aims to validate a smartphone-based pain assessment tool that patients can access at home.

DETAILED DESCRIPTION:
1. Purpose:

   The purpose of this study is to establish whether the Panda versions of the 100mm VAS (Visual Analogue Scale) and NRS-11 (Numeric Rating Scale) agree adequately with and can therefore be used in lieu of already validated paper versions of these scales for the evaluation of post-operative pain in adults. The Panda versions of the pain assessment scales have been condensed in size onto an iPod Touch screen but otherwise appear the same as traditional paper versions.
2. Hypothesis:

   There are no significant differences in the failure rates in obtaining pain scores and the pain scores obtained using Panda versions of the 100mm VAS and NRS-11 compared to the traditional paper versions.
3. Justification:

   The management of acute post-operative pain has a profound impact on a patient's short- and long-term wellbeing. Studies have shown that up to 70-80% of patients experience pain after surgery, with the majority reporting moderate, severe or extreme pain at some point. Ineffective pain management can increase the risk of venous thromboembolism, ischemic heart disease, pneumonia, poor wound healing , insomnia, anxiety and chronic post surgical pain (CPSP). The management of postoperative pain after patients leave hospital is especially inadequate, with more patients reporting pain after discharge than before. Although peripheral nerve blocks (PNB) have demonstrated benefit in reducing immediate/in-hospital postoperative pain compared to general anesthesia (GA), this benefit is not sustained after patients are discharged. In fact, more patients who received PNB report their pain as "severe", "excruciating" or "extreme" and seek medical attention after leaving hospital, than those who were under GA. The nociceptive barrage after the signal blockade by regional anesthesia wears off can theoretically lead to hyperalgesia, and the substantial increase in acute pain over a period of hours can be highly traumatic for patients. In order to minimize this effect, patients are often advised to begin the titration of their oral analgesics prior to the resolution of their nerve blocks, often when they do not feel much pain yet. Potential barriers encountered during this process can include the lack of incentive to begin analgesics in the presence of residual nociceptive blockade, the difficulty of titrating medications away from the direct supervision of medical professionals, and the fear of medication overdose. Therefore, detailed, easily comprehensible and patient specific pain management instructions need to be provided as a part of the discharge plan in order to facilitate patient compliance.

   The first step involves developing a practical tool that allows for the accurate and reliable assessment and recording of pain severity that patients can use from home. Pain is defined as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage". It is a highly individual experience. Therefore, self-report is considered the gold standard for pain assessment, with the Verbal Rating Scale (VRS), Visual Analogue Scale (VAS) and Numeric Rating Scale (NRS) being the three most validated self-report scales in adults. The VAS-100mm is a 100mm line with the anchoring words "no pain" and "worst imaginable pain" at the bottom and top, respectively. The NRS-11 is a line marked with numbers from 0 to 10 at even intervals, with the anchoring words "no pain" and "worst pain imaginable" at 0 and 10, respectively. Digital versions of pain scales that can be downloaded onto a smartphone have been found to be comparable to traditional paper versions in terms of their ability to measure pain. In addition to being portable and accessible, the digitization of pain assessments have the potential to reduce human errors that could occur during scoring and data recording. Furthermore, there is growing evidence that smartphone applications (apps) have the potential to improve compliance with disease and medication management by motivating patients to be involved in their own care. These properties make them promising tools for the management of postsurgical pain at home. The smartphone application "Panda" (Pain Assessment using a Novel Digital Application) developed by the British Columbia Children's Hospital (BCCH) Pediatric Anesthesia Research Team (PART), includes digital versions of the Faces Pain Scale - Revised (FPS-R) and Color Analog Scale (CAS), and has been validated in the pediatric population. Because the 100mm VAS and the 11-point NRS have been studied specifically in adults as tools for the evaluation of postoperative pain, the app will be modified to include these two scales to better suit this population.
4. Objectives:

   Panda will be compared against the traditional versions for both the NRS-11 and 100mm VAS to analyse the following endpoints:
   * Agreement between the two measures - the Panda score and the "traditional" score.
   * Practicality: difference in failure rates in obtaining pain scores from Panda compared with the "traditional" methods
5. Research design:

   This is an observational, randomized, cross-over controlled, open trial.
6. Statistical analysis:

   * Practicality: Chi-squared tests will be used to assess the difference in failure rates in obtaining pain scores from Panda compared with the "traditional" methods
   * Agreement: an interval approach described by Bland & Altman will be used to calculate the agreement between the the Panda scores and the 'traditional' scores.

Sample size: There will be 2 study groups- the 100mm VAS and NRS-11 groups. Each group will contain 2 subgroups - ages >18 to < 60 years and ≥60 to ≤ 75 years. The required sample of 32 patients per subgroup has been calculated on the basis of Liao's proposed sample size calculation for an agreement study based on the Bland-Altman interval method, setting the discordance rate (α) = 0.05 and the tolerance probability (β) = 80%. 160 patients will be recruited to allow for any unplanned gaps in data collection, patients withdrawing from the study and other exclusions

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 75
* ASA status I-III
* Undergoing a procedure with anticipated post-surgical pain

Exclusion Criteria:

* Undergoing eye surgery
* Significant cognitive impairment or neurological injury
* Psychomotor dysfunction
* Visual impairment
* Admission to the Intensive Care Unit.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
Scale Agreement at Time Zero: Difference between two modes of administration of the visual analogue scale (VAS-100) | Time zero took place in the postanesthesia care unit (PACU) within 15 minutes of emergence from general anesthesia or procedural sedation, after being deemed appropriate to assess by the bedside nurse
  Comparison of two modes of administration of the VAS-100 (paper and smartphone). Investigators will report only the mean difference in pain intensity between the two scales.Both scales will be administered adjacently, the order will be randomly assigned.
Scale Agreement at Time Zero: Difference between two modes of administration of the numeric rating scale (NRS-11) | Time zero took place in the postanesthesia care unit (PACU) within 15 minutes of emergence from general anesthesia or procedural sedation, after being deemed appropriate to assess by the bedside nurse
  Comparison of two modes of administration of the NRS-11 (paper and smartphone). Investigators will report only the mean difference in pain intensity between the two scales.Both scales will be administered adjacently, the order will be randomly assigned.
Scale Agreement at Time One: Difference between two modes of administration of the visual analogue scale (VAS-100) | Time One occurred when the patient met the postanesthesia care unit (PACU) discharge criteria as per institutional protocol, modified from PADSS (post anesthesia discharge scoring system), with minimum score 9/10. Up to 72 hours.
  Comparison of two modes of administration of the VAS-100 (paper and smartphone). Investigators will report only the mean difference in pain intensity between the two scales.Both scales will be administered adjacently, the order will be randomly assigned.
Scale Agreement at Time One: Difference between two modes of administration of the numeric rating scale (NRS-11) | Time One occurred when the patient met the postanesthesia care unit (PACU) discharge criteria as per institutional protocol, modified from PADSS (post anesthesia discharge scoring system), with minimum score 9/10. Up to 72 hours.
  Comparison of two modes of administration of the NRS-11 (paper and smartphone). Investigators will report only the mean difference in pain intensity between the two scales.Both scales will be administered adjacently, the order will be randomly assigned.

SECONDARY OUTCOMES:
Preference of smartphone app or traditional visual analogue scale (VAS-100) | Before PACU discharge, the subjects were asked whether they preferred the Smartphone app, the original tool, or had no preference.
  The participants were asked whether they preferred the Smartphone app, the original tool, or had no preference.
Preference of smartphone app or traditional numeric rating scale (NRS-11) | Before PACU discharge, the subjects were asked whether they preferred the Smartphone app, the original tool, or had no preference.
  The participants were asked whether they preferred the Smartphone app, the original tool, or had no preference.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Yarnold, MD, Principal Investigator — Providence Health & Services
Locations (2):
- Canada (2):
  - Mount Saint Joseph Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sun T, West N, Ansermino JM, Montgomery CJ, Myers D, Dunsmuir D, Lauder GR, von Baeyer CL. A smartphone version of the Faces Pain Scale-Revised and the Color Analog Scale for postoperative pain assessment in children. Paediatr Anaesth. 2015 Dec;25(12):1264-73. doi: 10.1111/pan.12790. PMID 26507916
- [Background] Sunderland S, Yarnold CH, Head SJ, Osborn JA, Purssell A, Peel JK, Schwarz SK. Regional Versus General Anesthesia and the Incidence of Unplanned Health Care Resource Utilization for Postoperative Pain After Wrist Fracture Surgery: Results From a Retrospective Quality Improvement Project. Reg Anesth Pain Med. 2016 Jan-Feb;41(1):22-7. doi: 10.1097/AAP.0000000000000325. PMID 26650425